CLINICAL TRIAL: NCT03806322
Title: A Better Way to Decrease Knee Swelling in Patients With Knee Osteoarthritis: A Single-Blind Randomized Controlled Trial
Brief Title: A Better Way to Decrease Knee Swelling in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MU2019VT
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold-pack Group (Experimental): One group received ultrasound, transcutaneous electrical nerve stimulation, electrical stimulation, exercise, and cold packs
  Interventions: Other: Cold-pack
- Intermittent Pneumatic Compression (Experimental): The second group received ultrasound, transcutaneous electrical nerve stimulation, electrical stimulation, exercise, and intermittent pneumatic compression
  Interventions: Other: Intermittent Pneumatic Compression

INTERVENTIONS:
Other: Intermittent Pneumatic Compression — The group received ultrasound, transcutaneous electrical nerve stimulation, electrical stimulation, exercise, and intermittent pneumatic compression.
  Arms: Intermittent Pneumatic Compression
Other: Cold-pack — The group received ultrasound, transcutaneous electrical nerve stimulation, electrical stimulation, exercise, and cold packs.
  Arms: Cold-pack Group

SUMMARY:
In this study, we compared the effects of intermittent pneumatic compression along with conventional treatment and cold-pack treatment along with conventional treatment on clinical outcomes in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with knee OA according to the criteria of the American College of Rheumatology (ACR), and were considered as stage 2 and 3 according to Kellgren-Lawrence criteria.

Exclusion Criteria:

Exclusion criteria were previous knee surgery, malignancy, circulation disorder, and conditions preventing exercise or causing muscle weakness, pregnancy, diagnosis of mental disorder, scar tissue, or metal implants.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2012-05-31 (Actual); Study Completion 2012-06-01 (Actual)

PRIMARY OUTCOMES:
Knee Swelling | 3 minutes
  Knee swelling was measured with a tape measure.
Pain Intensity | 3 minutes
  A Visual Analogue Scale was used to measure pain intensity.

SECONDARY OUTCOMES:
Range of Motion | 3 minutes
  A universal goniometer was used to measure range of knee flexion.
Muscle Strength | 10 minutes
  A digital dynamometer (J-TECH Power Track II Commander, USA) was used to measure quadriceps femoris and hamstring muscle strength.
Functional Status | 10 minutes
  The Western Ontario and McMaster Universities Arthritis (WOMAC) Index was used to evaluate pain, stiffness and physical function.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sari Z, Aydogdu O, Demirbuken I, Yurdalan SU, Polat MG. A Better Way to Decrease Knee Swelling in Patients with Knee Osteoarthritis: A Single-Blind Randomised Controlled Trial. Pain Res Manag. 2019 May 2;2019:8514808. doi: 10.1155/2019/8514808. eCollection 2019. PMID 31191790